CLINICAL TRIAL: NCT04312854
Title: A Prospective Cohort Study of Idiopathic Retroperitoneal Fibrosis in China
Brief Title: A Prospective Cohort Study of IRPF in China
Acronym: IRPF
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Wen Zhang, Professor, Peking Union Medical College Hospital
Other Study IDs: IRPF-Cohort in China
Record Dates: First submitted 2020-01-17; First posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Idiopathic Retroperitoneal Fibrosis
Keywords: idiopathic retroperitoneal fibrosis; Registry; cohort study
MeSH Terms: conditions — Retroperitoneal Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — Blood samples(serum and plasma,with DNA)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

SUMMARY:
This is a cohort study to investigate the disease course and treatment response of patients with idiopathic retroperitoneal fibrosis（IRPF）.

Methods: All the patients fulfilling diagnostic criteria of IRPF would be enrolled around China. A online database system will been established.

Endpoints: The primary endpoint is to investigate the clinical manifestations of Chinese IRPF patients; the secondary endpoints including the demographic features,laboratory characteristics, immunological tests, imaging and pathological features, in addition, the treatment and prognosis of the disease.

DETAILED DESCRIPTION:
Idiopathic retroperitoneal fibrosis（IRPF） is a rare fibro-inflammatory disease that develops around the abdominal aorta and the iliac arteries, and spreads into the adjacent retroperitoneum, where it frequently causes ureteral obstruction and renal failure. The clinical phenotype of RPF is complex, because it can be associated with fibro-inflammatory disorders involving other organs, and often arises in patients with other autoimmune conditions.

This prospective cohort aims to study presentations of IRPF with laboratory findings and imagings throughout the disease course. Newly diagnosed IRPF patients will be recruited from all over the China.

Inclusion criteria: patients with definite, possible IRPF will be recruited.Definite IRPF must have the following characteristics: (1) The typical finding of Imaging shows retroperitoneal mass, surrounding the abdominal aorta and iliac arteries, with encasement of ureters and/or organ dysfunction; (2) Exclusion of disease progression after standard glucocorticoid treatment; and (3) histopathological findings shows a ﬁbrous tissue with signs of chronic inﬂammation. The inﬂammatory component is comprised of lymphocytes, plasma cells and macrophages. Neutrophils and granulomas are rare ﬁndings. Possible IRPF required (1) and (2), but without histopathological examination.

Exclusion criteria: patients with malignancy or other autoimmune diseases are excluded. Secondary forms of RPF related to drugs, infections, malignancies, Erdheim-Chester disease and IgG4-RD, need to be excluded.

The data will be uploaded through the platform of Chinese Rheumatology Information Platform. Demographic data, initial symptoms, disease duration, and physical examination, organ involvements, laboratory findings, radiological and pathological results, as well as treatment, side effects will be recorded.

This study was approved by the Medical Ethics Committee of PUMCH (Beijing, China). All patients will sign informed consent.

Statistical Analysis: All parameters are described in the standard summary statistics, including mean, standard deviation, minimum, and maximum. All statistical analyses will be performed by SPSS.

Endpoints: The primary endpoint is to investigate the organ involvements of Chinese IRPF patients. The secondary endpoints including the demographic features,laboratory characteristics, immunological tests, imaging and pathological features, in addition, the treatment and prognosis of the disease.

ELIGIBILITY:
Inclusion Criteria:

Males and females; 18-75 years old with informed consent; Patients diagnosed with definite or possible IRPF.

Exclusion Criteria:

Secondary forms of IRPF; Pregnant or Females planning to bear a child recently ; Concurrent severe and/or uncontrolled and/or unstable diseases; Patients with malignancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with newly diagnosed IRPF
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-01-17 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Organ involvements of Chinese IRPF patients | 5 years
  To calculate the percentage of organ involvements in at least 500 patients.

SECONDARY OUTCOMES:
Response rate of glucocorticoids and immunosuppressants on IRPF in China | 5 years
Relapse rate of IRPF patients in China | 5 years
The correlation between baseline disease activities and relapse rate. | 5 years
Ten-year survival rate of patients with IRPF in China. | 10 years
The imaging features of involved organs. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Wen Zhang, MD, Principal Investigator — Department of Rheumatology,Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes